CLINICAL TRIAL: NCT05920421
Title: Diaphragm Sparing Effect of Subomohyoid Block With Infraclavicular or Subscapularis Blocks in Comparison With Interscalen Block for Postoperative Analgesia in Shoulder Surgeries
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Zagazig University (Other Government)
Responsible Party: Principal Investigator, Emad Hamdy Mohamed Morsy, assistant lecturer of anethesia and surgical intensive care, Zagazig University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: #6024/5-4-2022
Record Dates: First submitted 2023-05-14; First posted 2023-06-27 (Actual); Last update posted 2026-01-02 (Actual); Status verified 2025-12

CONDITIONS: Shoulder Surgeries Operations

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- interscalen group (Placebo Comparator): (29) patients will receive an interscalene block before induction of general anaesthesia.
  Patients will receive 20 ml of bupivacaine 0.25 %+250 mg of magnesium sulphate.
  Interventions: Procedure: diaghragm affection by ultrasound before and after the blocks
- subomohyoid infracavicular group (Active Comparator): (29) patients will receive subomohyoid infraclavicular block before induction of general anesthesia. Patients will receive 20 ml of bupivacaine 0.25 %+250 mg of magnesium sulphate.
  Interventions: Procedure: diaghragm affection by ultrasound before and after the blocks
- subomohyoid subscapularis group (Active Comparator): (29) patients will receive subomohyoid subscapularis block before induction of general anesthesia. Patients will receive 20 mL of 0.25% bupivacaine + 250 mg of magnesium sulfate.
  Interventions: Procedure: diaghragm affection by ultrasound before and after the blocks

INTERVENTIONS:
Procedure: diaghragm affection by ultrasound before and after the blocks — the participant will assess diaphragm sparing in each block and evaluate effectiveness of infraclavicular subomohyoid blocks and subomohyoid subscapularis blocks according to intraoperative and postoperative analgesia and diaphragm affection and comparing them with interscalen and with each others

SUMMARY:
The gold standard for shoulder analgesia is the interscalene block (ISB), but it has its own share of disadvantages such as phrenic nerve block, recurrent laryngeal nerve involvement and Horner's syndrome may lead to patient discomfort .Others, such as intrathecal spread and systemic toxicity of local anesthetic, can have serious consequences.

Phrenic nerve injury is a common complication with regional anesthesia. Its either temporary with Transient Phrenic Nerve Palsy leading to hemidiaphragmatic paresis after interscalene block or other injections of local anesthetic in the neck .

Although studies of ISB have shown a reduction in the incidence in hemidiaphragmatic paralysis with low-volume ISB, the risk of phrenic paralysis is not completely eliminated.

To bypass this complication, distal block of the shoulder innervation is recommended such as subomohyoid infraclavicular and subomohyoid subscapularis blocks.

DETAILED DESCRIPTION:
Ultrasound has a significant role in recent anesthesia. It plays a significant role in detecting diaphragmatic mobility and detecting phrenic nerve palsy after regional anesthesia . the common and standard technique for shoulder analgesia is interscalen block. but it has its own complications like phrenic nerve palsy.

to bypass this complications ,several ways had been tried to overcome this complications.

in this study, the investigator compare between the standard interscalen block with distal blocks like infraclavicular subomohyoid block and subomohyoid subscapularis blocks according to diaghragm affection , duration of analgesia , side effects occured with blocks.

For infraclavicular subomohyoid block, the infraclavicular approach targets the posterior and lateral cords, thus anesthetizing the axillary nerve (which supplies the anterior and posterior shoulder joint), whereas the suprascapular nerve block done by blocking subomohyoid muscle anesthetizes the posterior shoulder.

For subscapularis subomohyoid block, subscapularis is done before subomohyoid block. Subscapularis block target subscapular nerve which arise from posterior cord and present on ventral surface of subscapularis muscle .

ELIGIBILITY:
Inclusion Criteria:

* Patient acceptance.
* ASA I and ASA II.
* Age 21-60 years old.
* Both gender.
* BMI < 35 Kg/m2.
* Accepted mental state of the patient.
* Elective Unilateral upper limb surgeries at the level of the shoulder.
* Time of surgery less than 2 hours

Exclusion Criteria:

* - Patient refusal.
* Peripheral neuropathy.
* Pathological coagulopathy.
* Infection at the injection site.
* Untreated pneumothorax.
* Disturbed conscious level.
* An allergy to local anesthetics used in this study

Ages: 21 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 87 (Actual)
Dates: Start 2023-07-20 (Actual); Primary Completion 2023-12-20 (Actual); Study Completion 2024-12-30 (Actual)

PRIMARY OUTCOMES:
Change is being assessed (Diaphragm excursion) | basal preoperatively , immediately postoperatively in the pacu and 6 hours postoperatively
  As shown before diaphragm excursion will be examined preoperative as basal measurement, immediately postoperative in the PACU and 6 hours postoperatively to detect diaghragm excursion.If ratio of post to pre-block is < 25% this means that phrenic nerve block is included.
Thickness fraction | basal preoperatively, immediately postoperatively in the PACU, and 6 hours postoperatively
  The percentage change in thickness between end expiration and peak inspiration. It was calculated as follows: (thickness at peak inspiration - thickness at end expiration/thickness at end expiration) ×100.

SECONDARY OUTCOMES:
Visual Analogue Scale (VAS) at different intervals within and between the studied groups | immediately postoperative in the PACU , 6 hours postoperatively up to 24 hour postoperatively
  The investigators ask the patient to estimate the degree of pain on a scale from 1 to 10 and ask the patient to report the degree of pain from 0 to 10, with 0 no pain to 10 worst pain.
Total pethidine consumption in 24 hours of the studied groups | 24 hours
  The investigator will calculate the total amount of pethidine consumed over a 24-hour period.
postoperative complication of the studied groups | 24 hours
  the investigator will record patients with complications from the blocks like hypoxemia with saturation <90% , bradycardia with heart rate <50, nausea and vomiting

CONTACTS AND LOCATIONS:
Locations (1):
- Emad Hamdy Mohamed Morsy, Zagazig, Sharqia Province, Egypt

IPD SHARING:
Plan to Share IPD: Yes
planned after completion of the study
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: after puplication of the study
Access Criteria: contact of principal investigator

REFERENCES:
- [Background] Dhir S, Sondekoppam RV, Sharma R, Ganapathy S, Athwal GS. A Comparison of Combined Suprascapular and Axillary Nerve Blocks to Interscalene Nerve Block for Analgesia in Arthroscopic Shoulder Surgery: An Equivalence Study. Reg Anesth Pain Med. 2016 Sep-Oct;41(5):564-71. doi: 10.1097/AAP.0000000000000436. PMID 27380105
- [Background] Battaglia PJ, Haun DW, Dooley K, Kettner NW. Sonographic measurement of the normal suprascapular nerve and omohyoid muscle. Man Ther. 2014 Apr;19(2):165-8. doi: 10.1016/j.math.2013.12.005. Epub 2013 Dec 27. PMID 24412231
- [Background] Musso D, Flohr-Madsen S, Meknas K, Wilsgaard T, Ytrebo LM, Klaastad O. A novel combination of peripheral nerve blocks for arthroscopic shoulder surgery. Acta Anaesthesiol Scand. 2017 Oct;61(9):1192-1202. doi: 10.1111/aas.12948. Epub 2017 Aug 4. PMID 28776638
- [Background] Bergmann L, Martini S, Kesselmeier M, Armbruster W, Notheisen T, Adamzik M, Eichholz R. Phrenic nerve block caused by interscalene brachial plexus block: breathing effects of different sites of injection. BMC Anesthesiol. 2016 Jul 29;16(1):45. doi: 10.1186/s12871-016-0218-x. PMID 27473162
- [Background] Panero AJ, Hirahara AM. A Guide to Ultrasound of the Shoulder, Part 2: The Diagnostic Evaluation. Am J Orthop (Belle Mead NJ). 2016 May-Jun;45(4):233-8. PMID 27327915
- [Background] Boon AJ, O'Gorman C. Ultrasound in the Assessment of Respiration. J Clin Neurophysiol. 2016 Apr;33(2):112-9. doi: 10.1097/WNP.0000000000000240. PMID 27035251
- [Background] Jensen MP, Chen C, Brugger AM. Interpretation of visual analog scale ratings and change scores: a reanalysis of two clinical trials of postoperative pain. J Pain. 2003 Sep;4(7):407-14. doi: 10.1016/s1526-5900(03)00716-8. PMID 14622683
- [Result] Aszmann OC, Dellon AL, Birely BT, McFarland EG. Innervation of the human shoulder joint and its implications for surgery. Clin Orthop Relat Res. 1996 Sep;(330):202-7. doi: 10.1097/00003086-199609000-00027. PMID 8804294